CLINICAL TRIAL: NCT05064020
Title: Bictegravir in the Elderly Living With HIV: Impact of Polypharmacy and Multimorbidity (BICEP)
Brief Title: Bictegravir in the Elderly Living With HIV (BICEP)
Status: Active, not recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Qing Ma, PharmD, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00003629
Record Dates: First submitted 2020-07-15; First posted 2021-10-01 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: HIV-1-infection
Keywords: HIV; Switch; Bictegravir; Drug-drug interaction; Polypharmacy; Elderly; Adherence; Quality of life
MeSH Terms: interventions — bictegravir; Emtricitabine; tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Polypharmacy: Polypharmacy: patient is using five or more medications will be considered polypharmacy.
  Subjects having polypharmacy condition with taking Elvitegravir/Cobicistat/Emtricitabine/Tenofovir/Alafenamide 150MG-150MG-200MG-10MG Oral Tablet [Genvoya] or Elevitegravir/Cobicistat/Emtricitabine/Tenofovir disoproxil fumarate 150MG-150MG-200MG-300MG Oral Tablet [Stribild] will switch to Bictegravir/Emtricitabine/Tenofovir Alafenamide 50 MG-200 MG-25 MG Oral Tablet [BIKTARVY]
  Interventions: Drug: Bictegravir/Emtricitabine/Tenofovir Alafenamide 50 MG-200 MG-25 MG Oral Tablet [BIKTARVY]
- Nonpolypharmacy: Nonpolypharmacy: patient is using less than five medications will be considered nonpolypharmacy
  Nonpolypharmacy Subjects taking Elvitegravir/Cobicistat/Emtricitabine/Tenofovir/Alafenamide 150MG-150MG-200MG-10MG Oral Tablet [Genvoya] or Elevitegravir/Cobicistat/Emtricitabine/Tenofovir disoproxil fumarate 150MG-150MG-200MG-300MG Oral Tablet [Stribild] will switch to Bictegravir/Emtricitabine/Tenofovir Alafenamide 50 MG-200 MG-25 MG Oral Tablet [BIKTARVY]
  Interventions: Drug: Bictegravir/Emtricitabine/Tenofovir Alafenamide 50 MG-200 MG-25 MG Oral Tablet [BIKTARVY]

INTERVENTIONS:
Drug: Bictegravir/Emtricitabine/Tenofovir Alafenamide 50 MG-200 MG-25 MG Oral Tablet [BIKTARVY] — Administer BIC/FTC/TAF 50/200/25 mg tablet by mouth once a day from day 1 to168.
  Other Names: Biktarvy; BIC/FTC/TAF

SUMMARY:
This is a prospective, open-label, single center, post-approval and post-marketing study. Current national guideline recommends an integrase strand inhibitors (INSTI) in combination with two nucleoside reverse transcriptase inhibitors (NRTIs) as standard of therapy for HIV-1 infected patients. INSTI-based regimen may require a potent CYP3A inhibitor such as cobicistat to increase INSTI's plasma concentration and prolongs half-life. However, co-administration with a CYP3A inhibitor may increase the risk of drug-drug interactions. A novel INSTI, bictegravir, does not need a booster for pharmacokinetic enhancement.

Hypothesis: switching HIV-1 infected patients from booster containing regimen to bictegravir based regimen would decrease the risk of drug-drug interactions caused by a booster and improve quality of life and adherence.

DETAILED DESCRIPTION:
Antiretroviral treatment consisting of integrase strand inhibitors (INSTI) in combination with two nucleoside reverse transcriptase inhibitors (NRTIs) has become the standard of therapy for HIV-1 infected patients (2017 DHHS Guidelines). The development and advancement of such therapy have resulted in improved prognosis, allowing a larger proportion of patients in United States (> 50%) with HIV-1 infection to be 50 years of age or older, which is defined by the CDC as "older adults". A novel INSTI, bictegravir (BIC), has been recently approved by FDA, available in a fixed dose combination with emtricitabine (FTC) and tenofovir alafenamide (TAF) as a novel single-tablet regimen (STR), BIKTARVY®. Similar to other INSTI, BIC prevents HIV replication by inhibiting HIV integration into the host cell. In vitro studies have shown its selectivity against HIV-1 infected cells with a low cytotoxic profile.

Elvitegravir, boosted with cobicistat, is currently available as part of a single-tablet formulation with FTC and TAF (GenvoyaTM) or with FTC and TDF (StribildTM). Unlike ritonavir, cobicistat has no antiretroviral activity, but has potent inhibitory effects on CYP3A44. Elvitegravir is primarily metabolized by CYP3A4 and its co-administration with cobicistat boosts elvitegravir plasma concentration and prolongs its half-life4. Concurrent use of a potent CYP3A4 inhibitor, e.g., cobicistat, with medications that are metabolized by CYP3A4 can significantly increase the risk of drug-drug interactions. With an increase in the average survivability age of HIV-infected patients, chances of polypharmacy due to multimorbidity, a term used to define the presence of two or more concurrent chronic medical conditions, increases. Two studies have demonstrated that older HIV+ individuals engaged in polypharmacy are more likely to experience potential drug-drug interactions (PDDI). Many chronic medications such as antidepressants, HMG-CoA reductase inhibitors (statins), and cardiovascular medications are metabolized by CYP3A4. Concurrent administration of these medications with GenvoyaTM and StribildTMcan lead to increases in PDDI. Such interactions can result in more adverse drug reactions, drug-related toxicity of narrow therapeutic index drugs, and variations in the efficacy of concurrent medications. However, unlike elvitegravir, BIC does not require a booster such as cobicistat for pharmacokinetic enhancement. Its use can result in reductions in PDDI caused by cobicistat in adults with polypharmacy. This can improve quality of life in general, adherence and can directly avoid DDI-related adverse effects.

Although antiretroviral therapy (ART), when used concurrently with certain medications, has an increased risk of PDDI, studies have suggested a low DDI profile of BIC. In this study, such benefits of bictegravir will be assessed through the evaluation of polypharmacy, PDDI, health-related quality of life, and adherence of HIV-infected subjects.

BIC/FTC/TAF related adverse drug events are possible in the study. Due to BIC's recent FDA approval, a comprehensive list on the possible adverse drug events has become available. Common side effects reported in clinical phase II and phase III studies include diarrhea, nausea, and headache. Serious adverse events, including lactic acidosis, severe hepatomegaly have been reported with nucleoside reverse transcriptase inhibitors, but are uncommon. The standard regimen of BIC/FTC/TAF will be used; if a regimen change occurs, participation in the study will be discontinued. Participants will be carefully screened and those with pre-conditions, such as morbid obesity, hepatitis B virus, hepatitis C virus co-infection will be documented in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals > 18 years of age.
* Able and willing to provide informed/signed consent.
* Presence of HIV-1 infection as documented by a licensed ELISA test kit and confirmed by Western blot or HIV RNA.
* Current antiretroviral therapy, Genvoya or Stribild for HIV-1 infection.
* At least 1 or more concurrent prescription medication.
* HIV VL < 50 for over 6 months, no current OI, no cancers

Exclusion Criteria:

* Use of drugs of abuse or alcohol which would interfere with adherence or completion of this study.
* Current antiretroviral therapy other than GenvoyaTM or StribildTM for HIV-1 infection.
* Pregnancy or breast-feeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to study entry and day of entry.
* Chronic, severe, or other medical conditions that, in the opinion of the investigator, would interfere with the subject's ability to participate in the protocol.
* Use of prohibited protocol-specified drugs, prescription or over-the-counter medication (see Section 6.4.2) within 14 days prior to study entry.
* Moderate or severe cognitive impairment by history that, in the opinion of the investigator, would interfere with the subject's ability to participate in the protocol
* Laboratory parameters documented within 21 days prior to study entry that would increase the risk for adverse events:

  1. Hemoglobin < 12.5 g/dL for men; < 11.5 g/dL for women;
  2. Platelet count < 100,000 platelets/mm 3;
  3. AST (SGOT) or ALT (SGPT) > 1.5 x the upper limit of normal (ULN);
  4. Estimated GFR < 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals > 18 years of age with HIV-1, currently on antiretroviral therapy, Genvoya or Stribild, at least 1 or more concurrent prescription medication and HIV viral load < 50 c/ml for over 6 months, no current OI, no cancers
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Potential Drug Drug Interaction (PDDI) | week 1 to week 24
  From week 1 to week 24 the study will assess PDDI and concurrent medications

SECONDARY OUTCOMES:
Adherence | Baseline, week 4, week 8, week 12 and week 24
  Study team will evaluate patient adherence
Lipid panel changes | Baseline and week 24
  Lipid panel including total cholesterol, low density lipoprotein, high density lipoprotein, and triglyceride, will be monitored at baseline and week 24
Blood pressure changes | Baseline and week 24
  Blood pressure will be monitored at baseline and week 24
Blood glucose changes | Baseline and week 24
  Blood glucose will be monitored at baseline and week 24
Health related quality of life | Baseline, week 12 and week 24
  Health related quality of life will be evaluated based on HIV Symptom Index (range 0-80, lower scores suggest better quality of life)
Neurocognitive impairment | Baseline, week 12 and week 24
  Neurocognitive impairment will be evaluated using Montreal Cognitive Assessment (MoCA) at baseline, week 12 and week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Ma, PharmD, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Evergreen Health, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified IPD only.
Time Frame: The data will be summarized and presented in the conferences and scientific journals.
Access Criteria: Please contact the principal investigator for an access to IPD.

REFERENCES:
- [Background] Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, Girard PM, Brar I, Daar ES, Wohl D, Rockstroh J, Wei X, Custodio J, White K, Martin H, Cheng A, Quirk E. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2063-2072. doi: 10.1016/S0140-6736(17)32299-7. Epub 2017 Aug 31. PMID 28867497
- [Background] Gleason LJ, Luque AE, Shah K. Polypharmacy in the HIV-infected older adult population. Clin Interv Aging. 2013;8:749-63. doi: 10.2147/CIA.S37738. Epub 2013 Jun 21. PMID 23818773
- [Background] Tsiang M, Jones GS, Goldsmith J, Mulato A, Hansen D, Kan E, Tsai L, Bam RA, Stepan G, Stray KM, Niedziela-Majka A, Yant SR, Yu H, Kukolj G, Cihlar T, Lazerwith SE, White KL, Jin H. Antiviral Activity of Bictegravir (GS-9883), a Novel Potent HIV-1 Integrase Strand Transfer Inhibitor with an Improved Resistance Profile. Antimicrob Agents Chemother. 2016 Nov 21;60(12):7086-7097. doi: 10.1128/AAC.01474-16. Print 2016 Dec. PMID 27645238
- [Background] Tseng A, Hughes CA, Wu J, Seet J, Phillips EJ. Cobicistat Versus Ritonavir: Similar Pharmacokinetic Enhancers But Some Important Differences. Ann Pharmacother. 2017 Nov;51(11):1008-1022. doi: 10.1177/1060028017717018. Epub 2017 Jun 19. PMID 28627229
- [Background] van den Akker M, Buntinx F, Metsemakers JF, Roos S, Knottnerus JA. Multimorbidity in general practice: prevalence, incidence, and determinants of co-occurring chronic and recurrent diseases. J Clin Epidemiol. 1998 May;51(5):367-75. doi: 10.1016/s0895-4356(97)00306-5. PMID 9619963
- [Background] Tseng A, Szadkowski L, Walmsley S, Salit I, Raboud J. Association of age with polypharmacy and risk of drug interactions with antiretroviral medications in HIV-positive patients. Ann Pharmacother. 2013 Nov;47(11):1429-39. doi: 10.1177/1060028013504075. PMID 24285760
- [Background] Sax PE, DeJesus E, Crofoot G, Ward D, Benson P, Dretler R, Mills A, Brinson C, Peloquin J, Wei X, White K, Cheng A, Martin H, Quirk E. Bictegravir versus dolutegravir, each with emtricitabine and tenofovir alafenamide, for initial treatment of HIV-1 infection: a randomised, double-blind, phase 2 trial. Lancet HIV. 2017 Apr;4(4):e154-e160. doi: 10.1016/S2352-3018(17)30016-4. Epub 2017 Feb 15. PMID 28219610
- [Background] Marzolini C, Back D, Weber R, Furrer H, Cavassini M, Calmy A, Vernazza P, Bernasconi E, Khoo S, Battegay M, Elzi L; Swiss HIV Cohort Study Members. Ageing with HIV: medication use and risk for potential drug-drug interactions. J Antimicrob Chemother. 2011 Sep;66(9):2107-11. doi: 10.1093/jac/dkr248. Epub 2011 Jun 16. PMID 21680580
- [Background] Mrus JM, Leonard AC, Yi MS, Sherman SN, Fultz SL, Justice AC, Tsevat J. Health-related quality of life in veterans and nonveterans with HIV/AIDS. J Gen Intern Med. 2006 Dec;21 Suppl 5(Suppl 5):S39-47. doi: 10.1111/j.1525-1497.2006.00644.x. PMID 17083499
- [Background] Justice AC, Rabeneck L, Hays RD, Wu AW, Bozzette SA. Sensitivity, specificity, reliability, and clinical validity of provider-reported symptoms: a comparison with self-reported symptoms. Outcomes Committee of the AIDS Clinical Trials Group. J Acquir Immune Defic Syndr. 1999 Jun 1;21(2):126-33. PMID 10360804
- [Background] Sax PE, Pozniak A, Arribas J, et al. Phase 3 randomized, controlled, clinical trial of bictegravir coformulated with FTC/TAF in a fixed-dose combination vs dolutegravir + FTC/TAF in treatment-naïve HIV-1-positive adults: Week 48 results. International AIDS Society (IAS) Conference on HIV Science; July 23-26, 2017; Paris, France. Levin: Conference reports for National AIDS Treatment Advocacy Project (NATAP); 2017.
- [Background] Horn JR, Hansten PD, Chan LN. Proposal for a new tool to evaluate drug interaction cases. Ann Pharmacother. 2007 Apr;41(4):674-80. doi: 10.1345/aph.1H423. Epub 2007 Mar 27. PMID 17389673
- [Background] Letendre SL, Ellis RJ, Ances BM, McCutchan JA. Neurologic complications of HIV disease and their treatment. Top HIV Med. 2010 Apr-May;18(2):45-55. PMID 20516524
- [Background] Ancuta P, Kamat A, Kunstman KJ, Kim EY, Autissier P, Wurcel A, Zaman T, Stone D, Mefford M, Morgello S, Singer EJ, Wolinsky SM, Gabuzda D. Microbial translocation is associated with increased monocyte activation and dementia in AIDS patients. PLoS One. 2008 Jun 25;3(6):e2516. doi: 10.1371/journal.pone.0002516. PMID 18575590
- See also: The link to the Citation that didn't find a PubMed ID — http://www.natap.org/2017/IAS/IAS_39.htm
- See also: The information related to Biktarvy package insert — https://www.biktarvyhcp.com/dosing-administration/dosing

DOCUMENTS (1):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05064020/Prot_000.pdf